CLINICAL TRIAL: NCT03116555
Title: A Prospective, Multicenter Clinical Study of Apatinib Plus Irinotecan as Second-line Treatment in Locally Advanced or Metastatic Gastric or Gastroesophageal Junctional Adenocarcinoma
Brief Title: Apatinib Plus Irinotecan as Second-line Treatment in AGC or EGJA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Shengjing Hospital (Other); General Hospital of Shenyang Military Region (Other); The People's Hospital of Liaoning Province (Other); Anshan Tumor Hospital (Other); Benxi Cental Hospital (Other); Liaoyang Central Hospital (Other); The Affiliated Tumor Hospital of Harbin Medical University (Unknown); The Second Affiliated Hospital of Harbin Medical University (Other); Panjin Central Hospital (Other); Jilin University Sino-Japanese Friendship Hospital (Unknown); The First Hospital of Jilin University (Other); Liaoyang Petrochemical General Hospital (Unknown)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology，The First Hospital of China Medical University, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOG0103
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Gastric Adenocarcinoma
Keywords: Apatinib; Irinotecan; Second-line; Metastatic Gastric Adenocarcinoma
MeSH Terms: interventions — apatinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan plus apatinib (Experimental): Irinotecan: 180mg/m2, ivgtt,given on the first day; Apatinib: initial dose: 250mg,oral,once a day, after meal ( try to take the medicine at the same time each day).
  Repeat the therapeutic schedule every 3 weeks till progressive disease or intolerable toxicities.
  Interventions: Drug: Apatinib; Drug: Irinotecan

INTERVENTIONS:
Drug: Apatinib — Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2).
Drug: Irinotecan — Irinotecan was used as second line treatment with AGC

SUMMARY:
This is a prospective, multicenter, single-group clinical study of Apatinib Plus Irinotecan as second-line treatment in locally advanced or metastatic gastric or gastroesophageal junctional adenocarcinoma.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-group clinical study of Apatinib Plus Irinotecan as second-line treatment in locally advanced or metastatic gastric or gastroesophageal junctional adenocarcinoma. Interventions: Irinotecan: 180mg/m2, ivgtt,given on the first day; Apatinib: initial dose: 250mg,oral,once a day, after meal ( try to take the medicine at the same time each day). Repeat the therapeutic schedule every 3 weeks till progressive disease or intolerable toxicities. Primary Outcome Measure: PFS. Secondary Outcome Measures: OS, ORR, DCR.

ELIGIBILITY:
Inclusion Criteria:

1. Age：18-70，female or male.
2. Pathologically diagnosed local advanced or metastatic stomach or gastroesophageal junction with adenocarcinoma, at least one measurable objective tumor lesion by spiral CT examination（according to RECIST 1.1）.
3. First-line application of fluorouracil-based chemotherapy failed (treatment failure definition: toxic side effects can not tolerate the progress of the disease during treatment or recurrence after treatment); Note:(1) Time of first-line treatment for subjects with advanced tumour must more than 1 cycles;(2) Adjuvant/neoadjuvant therapy was allowed; adjuvant/neoadjuvant therapy will be considered as a first-line treatment if disease recurrence during treatment or after less than 24 weeks.
4. UGT1A1*28(6/6) and *6(G/G) ,or UGT1A1*28(6/6) and *6(G/A),or UGT1A1*28(6/7) and *6(G/G).
5. ECOG performance status 0-1.
6. satisfactory main organ function，laboratory test must meet the following criteria: (1) blood routine examination standards to meet: A. HB≥90g/L; B. ANC≥1.5×109/L; C. PLT≥90×109/L; (2) biochemical tests to meet the following criteria: A. Total bilirubin≤1.5 times the upper limit of normal (ULN) B. ALT and AST≤2.5ULN; C. Serum Cr≤1ULN, endogenous creatinine clearance> 60ml/min (Cockcroft-Gault formula)
7. The international normalized ratio (INR) ≤ 1.5 and some prothrombin time (PPT or APTT) ≤ 1.5ULN within 7 days before participating.
8. Expected survival≥3 months;
9. Signed informed consent (ICF) before admission;
10. Women of childbearing age must undergo a pregnancy test (serum or urine) within 7 days prior to enrollment and have a negative result and are willing to use appropriate methods for contraception at 8 weeks after the trial and at the end of the last test. For men, contraception should be used for surgical sterilization, or agreed to use the appropriate method 8 weeks after the trial and the last given test drug.

Exclusion Criteria:

1. Hypersensitivity to apatinib, irinotecan or excipients.
2. More than one chemotherapy regimen was treated after progression of gastric cancer (except for adjuvant/neoadjuvant chemotherapy with more than 24 weeks of clearance).
3. Prior exposure to irinotecan.
4. Prior exposure to irinotecan VEGFR inhibitors, such as apotinib, sorafenib, sunitinib.
5. Another primary tumor in patients, except for: systematically treatment non-melanoma skin cancer, effectively treatment cervical carcinoma in situ, or other effectively treatment tumors wtih no recurrence for more than 5 years.
6. Anti neoplastic cytotoxic drugs, biological drugs (such as monoclonal antibodies), immunotherapy (such as interleukin 2 or interferon), or other research drugs have been use within 4 weeks before participating.
7. Uncontrolled hypertention with systolic blood pressure> 140 mmHg or diastolic blood pressure> 90 mmHg, grade I or more coronary heart disease, grade I arrhythmia (including QTc interval: male> 450 ms, female> 470 ms) and grade I cardiac insufficiency.
8. Urine routine urinary protein ≥ ++, or 24 hours urine protein ≥ 1g.
9. Any toxicity more than 1 grade(according to CTCAE) caused by previous treatment, except hair loss.
10. Occasional artery/venous thrombosis events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism occurred within 12 months before participation;
11. Intestinal obstruction occurred 4 weeks before participation.
12. Patients who underwent major surgery 4 weeks prior to initiation of treatment. The patient must be cured from any major surgery.
13. Patients who are considered to have a greater risk of medical care due to a serious, uncontrollable disease, non-metastatic systemic disease or active, uncontrollable infection. Some examples include, but not exclusively, uncontrolled ventricular arrhythmias, recent (3 months) myocardial infarction, uncontrollable epilepsy seizures, unstable spinal cord compression, superior vena cava syndrome, HRCT tips Bilateral interstitial lung disease or any mental illness that may obstruct informed consent.
14. Immunocompromised patients, for example, serological tests suggest that human immunodeficiency virus (HIV) is positive.
15. Pregnant or lactating women.
16. Have a variety of factors that affect oral medication (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.).
17. Patients with clear gastrointestinal bleeding tendencies. Including the following: there is black stool, hematemesis history in 2 months can not be grouped; For patient with fecal occult blood (+) and the primary tumor of the stomach tumor not surgical resected, if the center of the main investigators believe that there is possible occurrence of gastrointestinal bleeding,the patient can not be grouped.
18. Ascites or pleural effusion requiring clinical treatment of persistent.
19. A history or evidence of hereditary hemorrhagic physical or coagulopathy that increases the risk of bleeding.
20. With central nervous system metastasis with symptoms.
21. With Gilbert syndrome.
22. Participated in other drug clinical trials in four weeks.
23. Researchers believe that they are not suitable for inclusion.
24. Patients who had bone metastases and had undergone palliative radiotherapy (radiotherapy> 5% bone marrow area) within 4 weeks prior to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival [PFS] | 5-6 months
  Progression Free Survival

SECONDARY OUTCOMES:
Overall Survival [OS] | 12-15 months
  Overall Survival
Objective Response Rate [ORR] | 12-15 months
  Objective Response Rate
Disease Control Rate [DCR] | 12-15 months
  Disease Control Rate

OTHER OUTCOMES:
Incidence and Degree of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12-15 months
  Incidence and Degree of Treatment-Emergent Adverse Events
Performance Status [WHO-ECOG] | 12-15 months
  Performance Status
Quality of Life [WHO-QOL] | 12-15 months
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: YunPeng Liu, PhD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Result] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Result] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Result] Catalano V, Graziano F, Santini D, D'Emidio S, Baldelli AM, Rossi D, Vincenzi B, Giordani P, Alessandroni P, Testa E, Tonini G, Catalano G. Second-line chemotherapy for patients with advanced gastric cancer: who may benefit? Br J Cancer. 2008 Nov 4;99(9):1402-7. doi: 10.1038/sj.bjc.6604732. PMID 18971936
- [Result] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952
- [Result] Thuss-Patience PC, Kretzschmar A, Bichev D, Deist T, Hinke A, Breithaupt K, Dogan Y, Gebauer B, Schumacher G, Reichardt P. Survival advantage for irinotecan versus best supportive care as second-line chemotherapy in gastric cancer--a randomised phase III study of the Arbeitsgemeinschaft Internistische Onkologie (AIO). Eur J Cancer. 2011 Oct;47(15):2306-14. doi: 10.1016/j.ejca.2011.06.002. PMID 21742485